CLINICAL TRIAL: NCT00000742
Title: A Phase I Concentration-Controlled Trial to Assess the Safety, Tolerance, Pharmacokinetics and Development of Decreased HIV-1 Susceptibility to the Combination of Atevirdine Mesylate (U-87201E), Zidovudine (AZT), and Didanosine (ddI)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Upjohn (Industry); Glaxo Wellcome (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 199; 11175 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Didanosine; Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Antiviral Agents; Zidovudine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — atevirdine; Zidovudine; Didanosine

INTERVENTIONS:
Drug: Atevirdine mesylate
Drug: Zidovudine
Drug: Didanosine

SUMMARY:
Part I: To determine the pharmacokinetic dose for atevirdine mesylate ( U-87201E ) when used in combination with zidovudine ( AZT ). To determine the pharmacokinetic profiles of U-87201E and AZT over a 12-week period.

Part II: To determine whether or not decreased viral susceptibility to U-87201E develops when the drug is administered concomitantly with AZT for 12 weeks.

Part III: To evaluate the pharmacokinetic effects of ddI/AZT/U-87201E therapy and to assess changes in viral susceptibility to U-87201E.

Interest exists in the development of antiretroviral agents that possess different mechanisms of action from nucleoside analogs such as AZT. U-87201E is a non-nucleoside reverse transcriptase (RT) inhibitor that has demonstrated activity against HIV-1; however, an emerging characteristic of non-nucleoside RT inhibitors is the development of rapid resistance to HIV isolates. Whether this resistance can be prevented in the presence of nucleoside analogs such as AZT and ddI has yet to be determined.

DETAILED DESCRIPTION:
Interest exists in the development of antiretroviral agents that possess different mechanisms of action from nucleoside analogs such as AZT. U-87201E is a non-nucleoside reverse transcriptase (RT) inhibitor that has demonstrated activity against HIV-1; however, an emerging characteristic of non-nucleoside RT inhibitors is the development of rapid resistance to HIV isolates. Whether this resistance can be prevented in the presence of nucleoside analogs such as AZT and ddI has yet to be determined.

Part I: Five male patients enter a pharmacokinetic concentration-controlled trial of U-87201E plus zidovudine at the University of Rochester site only. A target plasma concentration range at trough for U-87201E will be determined. Pharmacokinetic monitoring continues for 7 days or until the desired dose regimen has been determined. The five patients may be eligible to continue in Part II of the study to complete a total of 12 weeks of therapy.

Part II: At least 10 male patients (all sites eligible) in addition to the five patients from Part I receive doses of U-87201E as determined by Part I and AZT at the same dose as in Part I. Therapy is administered for 12 weeks. Patients with no decreased viral susceptibility to U-87201E after 6 weeks may be offered an extension to 24 or more weeks of therapy. Patients are followed weekly for 8 weeks and every other week thereafter until the end of the study.

Part III: At least eight patients who have received 24 weeks of U-87201E/AZT have ddI added to the regimen for 12 additional weeks.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* PCP prophylaxis with aerosolized pentamidine, trimethoprim / sulfamethoxazole or dapsone.
* Clotrimazole troches or nystatin oral suspension for oral candidiasis.
* Acyclovir (up to 1000 mg/day) for herpes lesions.

Patients must have:

* HIV infection documented by serologic tests or HIV culture OR prior diagnosis of AIDS by established CDC criteria.
* CD4 counts = or < 500 cells/mm3 on two evaluations.

Part II only:

* No prior therapy with antiretroviral or immunomodulating agents (e.g., AZT, ddI, ddC, interferon).

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms and conditions are excluded:

* Acute medical problems at time of study entry (including active opportunistic infections such as active cryptococcosis, Pneumocystis carinii, herpes zoster, histoplasmosis, or CMV, or nonopportunistic diseases including liver disease, renal disease, orthostatic hypotension, hypertension, lymphoma).
* Current diagnosis of malignancy for which systemic therapy would be required during the study.

Concurrent Medication:

Excluded:

* Any other investigational drugs.
* Phenobarbital, phenytoin, ketoconazole, rifampin, cimetidine, beta blockers, chronic anti-acid therapy, antiarrhythmic agents or other medications known to affect cardiac conduction or seizure threshold.
* Cytotoxic chemotherapy.

Patients with the following prior conditions are excluded:

* History of cardiovascular disease including conduction disturbances, arrhythmias, atherosclerotic heart disease, or valvular heart disease.
* History of CNS disease such as seizure disorder, AIDS Dementia Complex, Progressive Multifocal Leukoencephalopathy, or any other active neurological disorder.
* History of active or chronic gastrointestinal disorders such as chronic diarrhea (> 4 weeks duration), constipation, unexplained abdominal pain (such as irritable bowel syndrome), or other GI motility disorders.
* History of hypercholesterolemia requiring medication or serum cholesterol = or > 300.

Part I patients only:

* History of inability to tolerate zidovudine (200 mg q 8 hours).

Part III patients only:

* History of pancreatitis or > grade 2 peripheral neuropathy.

Prior Medication:

Excluded:

* Cytotoxic chemotherapy within 1 month prior to study entry.

Part II only:

* prior therapy with antiretroviral or immunomodulatory agents (including but not limited to AZT, ddI, ddC, and interferon).

Current use of alcohol or illicit drugs.

Min Age: 13 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15
Dates: Study Completion 1993-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Reichman R, Study Chair
Locations (5):
- United States (5):
  - USC CRS, Los Angeles, California
  - Univ. of Miami AIDS CRS, Miami, Florida
  - Washington U CRS, St Louis, Missouri
  - Univ. of Rochester ACTG CRS, Rochester, New York
  - The Ohio State Univ. AIDS CRS, Columbus, Ohio

REFERENCES:
- [Background] Reichman RC, Morse GD, Demeter LM, Resnick L, Bassiakos Y, Fischl M, Para M, Powderly W, Leedom J, Greisberger C, et al. Phase I study of atevirdine, a nonnucleoside reverse transcriptase inhibitor, in combination with zidovudine for human immunodeficiency virus type 1 infection. ACTG 199 Study Team. J Infect Dis. 1995 Feb;171(2):297-304. doi: 10.1093/infdis/171.2.297. PMID 7531207
- [Background] Morse G, Fischl M, Leedom J, Batts D, Cox S, Reichman R. Atevirdine (ATV) pharmacokinetics (PK) and dosage requirements during a concentration-targeted (CT) phase I study (ACTG 199). Int Conf AIDS. 1993 Jun 6-11;9(1):477 (abstract no PO-B26-2050)
- [Background] Morse GD, Reichman RC, Fischl MA, Para M, Leedom J, Powderly W, Demeter LM, Resnick L, Bassiakos Y, Timpone J, Cox S, Batts D. Concentration-targeted phase I trials of atevirdine mesylate in patients with HIV infection: dosage requirements and pharmacokinetic studies. The ACTG 187 and 199 study teams. Antiviral Res. 2000 Jan;45(1):47-58. doi: 10.1016/s0166-3542(99)00073-x. PMID 10774589
- [Background] Reichman R, Fischl M, Para M, Powderly W, Timpone J, Bassiakos Y. Phase I study of atevirdine (ATV), a non-nucleoside reverse transcriptase inhibitor, given in combination with zidovudine (ZDV). The ACTG 199 Team. Int Conf AIDS. 1993 Jun 6-11;9(1):478 (abstract no PO-B26-2055)
- [Background] Demeter LM, Resnick L, Tarpley WG, Fischl M, Para M, Reichman RC. Prolonged sensitivity of HIV-1 isolates to atevirdine (ATV) in a phase 1 clinical trial of ATV and zidovudine (ZDV) (ACTG 199). The ACTG 199 Study Team. Int Conf AIDS. 1993 Jun 6-11;9(1):242 (abstract no PO-A26-0643)